CLINICAL TRIAL: NCT01135147
Title: Dietary Therapy for Obesity-related Sleep-disordered Breathing in Children
Brief Title: Obesity and Obstructive Sleep Apnea (OSA) in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Arnon Elizur, MD, Assaf Harofeh Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 40/09
Record Dates: First submitted 2010-05-31; First posted 2010-06-02 (Estimated); Last update posted 2010-06-02 (Estimated); Status verified 2010-05

CONDITIONS: Obstructive Sleep Apnea; Obesity
MeSH Terms: conditions — Sleep Apnea, Obstructive; Obesity | interventions — Diet; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diet (Experimental): Patients treated with diet and physical therapy for the entire 6 months of the study
  Interventions: Behavioral: Diet
- Surgery (Active Comparator): Patients undergoing adenotonsillectomy at some point of the study period
  Interventions: Procedure: Surgery

INTERVENTIONS:
Behavioral: Diet — Dietary therapy and physical education
  Arms: Diet
Procedure: Surgery — Adenotonsillectomy along with diet and physical therapy
  Arms: Surgery

SUMMARY:
The goal of this research is to study the prevalence of sleep disordered breathing and associated morbidity in obese children and to examine the role of diet and physical activity in the treatment of sleep-disordered breathing in obese children.

DETAILED DESCRIPTION:
In a prospective cohort study, obese children will be recruited. After informed consent is obtained, all children will complete a standardized sleep questionnaire and a pediatric daily sleepiness scale questionnaire. All participants will undergo a complete physical examination, blood tests for lipid profile, liver enzymes, and Glucose and insulin will be obtained, and liver sonography will be performed to assess for the presence of fatty liver. Nasopharyngeal radiographs will be used to assess adenoidal size based on the method by Cohen and Konak. A standard in-laboratory, overnight polysomnography will be performed, within 2 weeks of enrollment to the study, in the sleep laboratory at Asaf Harofeh Medical Center. Children with severe obstructive sleep apnea, defined as apnea hypopnea index (AHI) > 15 will undergo adenotonsillectomy. All children will be referred for a dietary and physical education program. The first visit with the dietician will be considered day 1 of the study. Children will than be followed monthly by a dietician. After three months of follow-up, subjects will be divided into two groups. Group 1 will include all children who had AHI > 2 on the initial polysomnography (including children who underwent adenotonsillectomy for AHI > 15), and group 2 will consist of children who had AHI < 2 on the initial PSG. Children of group 2 will continue monthly dietary visits as before. Children from group 1 will undergo a second evaluation including questionnaires, laboratory blood tests, liver sonography, nasopharyngeal radiographs, and polysomnography. Children who demonstrate reduction in the AHI based on PSG will be offered to continue with dietary treatment alone. Children with no change in the AHI based on PSG will be offered to undergo adenotonsillectomy in addition to continued dietary management. All children will be followed for a total duration of six months. After six months, all children will be re-evaluated by questionnaires, blood tests, liver sonography, and nasopharyngeal radiographs. Polysomnography will be performed in all children who had an AHI > 2 on the second PSG.

ELIGIBILITY:
Inclusion Criteria:

* BMI at or above the 90th percentile

Exclusion Criteria:

* children with chronic lung or liver disease, mental retardation, syndromes (i.e. prader willi syndrome), endocrine abnormalities (hypothyroidism cushing), chronic medical treatment with oral steroids, or with anti-psychiatric or anti-convulsive medications

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2010-06; Primary Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Reduction in apnea hypopnea index (AHI) | 3, 6 months
  Repeat polysomnography to assess change in AHI following treatment

SECONDARY OUTCOMES:
Change in subjective complaints and sleepiness | 6 months
Change in lipid profile and liver enzymes | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Asaf Harofeh Medical Center, Ẕerifin, Israel